CLINICAL TRIAL: NCT03355183
Title: Determining the Number of Repetitions Specific to Angular Speed of 60°\ Second and 180°\ Second in Establishing Isokinetic Knee Evaluation Protocols
Brief Title: Determining the Number of Repetitions Specific Isokinetic Knee Evaluation Protocols
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 34
Record Dates: First submitted 2017-11-22; First posted 2017-11-28 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Sports Physical Therapy
Keywords: isokinetics; knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy athletes (Experimental): Muscular strength of healthy athletes who are not physically disabled and doing sports for 3 years as a professional will be measured by isokinetic dynamometer.
  Interventions: Other: Isokinetics

INTERVENTIONS:
Other: Isokinetics — Isokinetics, or accommodating resistance, is a form of exercise where a person provides a maximum muscle contraction against a resistance or lever arm, (isokinetic dynamometer) at a fixed speed through a given range of motion. This type of muscle action can be done either concentrically or eccentrically at the given joint.

SUMMARY:
The aim of this study is to determine the repetition numbers of the peak force value generated during isokinetic knee flexion and extensor movement evaluation at 60 and 180 °/ sec angular velocities and to identify the factors associated with this repetition.

DETAILED DESCRIPTION:
Individual evaluation in the field of health; is very important because it sets out the steps necessary for defining and improving the current situation. Evaluation of muscular strength is a key factor in sports to improve performance and determine the risk of injury. Thus, the training and training process that will optimize the performance of the athlete can be planned and necessary steps can be taken to prevent injuries. There are many methods to determine muscle strength, manual muscle testing and isokinetic evaluation are the most frequently used methods. Isokinetic evaluation provides the ability to objectively measure dynamic force. Potential injuries are avoided by providing effective and optimal loading of joints and muscles throughout the range of motion. With isokinetic dynamometry, it can measure and amplify at high speed with maximal contraction using muscle function at full speed over the entire range of motion. With this method, it is possible to assess the strength of the muscles of the joint movements in the agonist (the group performing the movement as a primer) and the antagonist (the muscle group controlling the movement in the movement) during all reciprocal movements. One of the most important values of this evaluation is the peak torque, the maximum force. The peak torque value is influenced by many internal factors such as the environmental factors, the adaptation of the isokinetic instrument to the person, as well as the internal factors of the person being assessed. One of the most important of the effective factors is to determine the appropriate number of repetitions. Isokinetic dynamometers offer the possibility to make various adjustments such as angular velocity, number of repetitions, the range of motion, the current state of the person. Therefore, the evaluator can determine the number of repetitions itself. Sufficient repeatability is required to allow the individual to create maximum force. However, too much repetition can cause fatigue in the individual as well as an additional workload in terms of time. There are many studies in the literature carried out with different repeat numbers at different angular velocities. The studies include protocols ranging from five repetitions to twenty repetitions with very different repeat numbers. Five repetitions may not be sufficient for the peak torque to appear, but twenty repetitions cause fatigue in the athlete and lead to loss of time. There is no standardized repeat number for isokinetic knee evaluation in the literature. The lack of consensus on the number of repetitions hampers the interpretation of the works. In our work, it will be determined how many times the athletes reached peak torque values. This will prevent future studies from carrying out an incorrect measurement without reaching the maximum peak force with a low number of repetitions, or having too many repetitions to include tougher, longer evaluations. Standardization of repeat numbers will make evaluation easier and more meaningful if it increases the objectivity of evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Do sports for at least 3 years
* To have physical and mental fitness to perform isokinetic evaluation
* Being a mid-level workout (2-4 times a week)
* Volunteer to participate in the work.

Exclusion Criteria:

* • Hip, knee, ankle and back injuries in the last year

  * Having undergone lower extremity surgery
  * Having obstructive conditions such as muscular shortening that would prevent the movement gap to be standardized for isokinetic evaluation
  * Having a discomfort to affect neuromuscular control
  * In the last 6 months, intraarticular injection has been applied to the knee joint

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 196 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Isokinetic muscle strength's | 1 month
  the repetetion numbers of the peak force value generated during isokinetic knee flexion and extensor movement evaluation at 60 and 180 ° / will be assested with ISOMED 2000 device

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt Üniversitesi, Ankara, Turkey (Türkiye)